CLINICAL TRIAL: NCT03699501
Title: Psychometric Validation of an Oral Health-related Scale for Quality of Life and Coping in People With Schizophrenia
Acronym: QUALITY BIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DENIS 2018
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Surveys and Questionnaires; Diagnosis, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Questionnaires; Procedure: Oral examination
- Voluntary patients
  Interventions: Other: Questionnaires; Procedure: Oral examination; Other: questionnaires (test-retest)

INTERVENTIONS:
Other: Questionnaires — * A validated oral health-related quality of life self-assessment questionnaire: the GOHAI
  * A validated oral health-related quality of life self-assessment questionnaire to be validated: SOHP
  * A validated depression scale: the Beck scale
  * A self-assessment questionnaire for oral health coping to be validated: the SCOOHP
  * A validated self-assessment questionnaire for coping: The Brief cope)
Procedure: Oral examination — * An evaluation of dental health using the CAO index
  * An evaluation of oral hygiene with the IHO-S index
Other: questionnaires (test-retest) — SCOOHP and SOHP questionnaires
  Groups: Voluntary patients

SUMMARY:
Schizophrenia is a severe and persistent psychological disorder affecting 0.7 to 1% of the world's population and 600,000 people in France. Schizophrenic patients are exposed to excess mortality and a life expectancy that is 10 to 15 years lower than the general population (excluding causes of suicide) and to numerous co-morbidities, including oral diseases.

To improve this public health problem, concrete action must be undertaken and evaluated in both quantitative and qualitative terms. While there are many quantitative indicators, there are no reliable and valid tools for the perceived oral health of these individuals in the context of their real and/or imagined world.

The results of a qualitative study previously carried out by our team (QUALITY Study: NCT02730832) made it possible to develop two hypothetical questionnaires for evaluating quality of life related to oral health, the Schizophrenia Oral Health Profile (SOHP), and a questionnaire for evaluating coping strategies with regard to oral health, the Schizophrenia Coping Oral Health Profile (SCOOHP).

However, before these questionnaires can be used in clinical practice, their psychometric properties must be validated.

ELIGIBILITY:
Inclusion Criteria:

* Adult person,
* Patients for whom a diagnosis of schizophrenia is defined according to ICD 10
* Person who has given his or her oral agreement to participate in the study, with the agreement of the tutor in the context of a tutorship,
* Managed in a Specialised Institution (University Hospital, Psychiatric hospital or Hospital), either in full hospitalisation or on an outpatient basis,
* Fluent use of the French language.

Exclusion Criteria:

* Psychiatrically unstable and delusional patients.
* Patients with cognitive abilities too impaired to participate in the study
* Individuals with no natural teeth
* Pregnant or breastfeeding women
* Patients not affiliated to the national health insurance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Managed in a Specialised Institution (University Hospital, Psychiatric hospital or Hospital), either in full hospitalisation or on an outpatient basis
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
reliability of scales (internal consistency) | through study completion, an average of 18 months
validity of scales (consistency of responses) | through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France